CLINICAL TRIAL: NCT05286073
Title: Assessment of Vertical Root Fracture Resistance of Endodontically Treated Teeth Instrumented by Single Endodontic Files
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Urooj Musheer, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB-1658/DUHS/Approval/2020/
Record Dates: First submitted 2022-02-04; First posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Vertical Fracture of Root of Tooth (Disorder)
Keywords: Hyflex EDM,F6 Sky Taper,One Shape

STUDY DESIGN:
Intervention Model Description: Samples were randomly divided in 4 groups. Random sampling was done with computer generated method. There were 3 working groups comprising of 22 canals and 1 negative control group having 22 canals.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hyflex EDm (Experimental): The canals were prepared and shaped with one file (25/~) and finished with 40/.04 using crown down technique. Torque controlled endodontic motor was used with a rotational speed of 500 rpm and torque of 2.5Ncm (25 Nm).
  Interventions: Procedure: Endodontic Root Canal Treatment
- F6 SkyTaper (Experimental): The canals were prepared and shaped with one file (25/~) and finished with 40/.04 using crown down technique. Torque controlled endodontic motor was used with a rotational speed of 500 rpm and torque of 2.5Ncm (25 Nm).
  Interventions: Procedure: Endodontic Root Canal Treatment
- One Shape (Experimental): Canals were prepared and shaped with single rotational file system One Shape with the sequence of Endoflare (12, 0.12), One G (18, 0.03) and One Shape (12.06) connected to endodontic motor with rotational speed of 400rpm and 4 Ncm torque as recommended by manufacturer.
  Interventions: Procedure: Endodontic Root Canal Treatment
- Control (No Intervention): In the control group, no endodontic instrumentation and shaping was done in the canals. Only the necrotic pulp tissue was extirpated from the canals with the help of barbed broaches and then the specimens were analyzed for fracture testing.

INTERVENTIONS:
Procedure: Endodontic Root Canal Treatment — Root canal shaping procedures were performed. Irrigation was done after each three pecks of endodontic file. After instrumentation (Groups 1-3), the canals were dried with sterile paper points. The dentinal walls were then coated with Sealapex. For vertical root fracture resistance testing, sample preparation was done in acrylic blocks. Then roots were coated with polyvinylsiloxane impression material. After that roots were inserted again into acrylic resin blocks. The acrylic blocks with the vertically aligned roots were mounted in the Instron testing machine. 0.5 mm diameter round tip stainless-steel rod was fixed to the universal testing machine. The universal testing machine was adjusted and vertical compressive force was applied at a crosshead speed of 1mm/min. The Instron tester applied a slowly increasing force, until the root fractured. The maximum amount of force necessary to fracture every sample was recorded in Newton (N).
  Arms: F6 SkyTaper; Hyflex EDm; One Shape

SUMMARY:
The purpose of this study is the assessment of vertical root fracture resistance of roots prepared with three different single endodontic rotary files in extracted human mandibular premolar roots.

DETAILED DESCRIPTION:
88 human extracted mandibular premolars will be selected. Teeth will be sectioned below cementoenamel junction to get 13mm from the apex of root. Roots will then be standardized according to buccolingual and mesiodistal widths and will be examined for fracture and craze lines. The roots will then be randomly divided into 3 experimental groups and 1 control group (n=22). Group 1 will be instrumented with Hyflex EDM. Group 2 will be instrumented with F6 Sky Taper. Group 3 will be instrumented with One Shape and Group 4 will be negative control group in which no instrumentation will be done. After performing rotary instrumentation, roots will then be obturated with respective GP and sealer. Samples will then be exposed to vertical load utilizing Universal Testing Machine till fracture occur which will be recorded in Newton(N).

ELIGIBILITY:
Inclusion Criteria:

* Extracted Human mandibular premolar canals that fulfill the following criteria were used.

  * permanent teeth
  * intact and fully formed apices
  * straight and single rooted canal
  * roots having similar diameter mesiodistally(2-4mm) and buccolingually(4-6mm)

Exclusion Criteria:

* Roots having following features were excluded;

  * root caries
  * roots with multiple canals
  * previous root canal treatment done
  * signs of calcification, internal and external root resorption
  * cracks
  * fracture lines
  * C-shaped canals
  * Vertical Root Fracture

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Vertical Root Fracture Resistance | 5 minutes
  The acrylic blocks with the vertically aligned roots were mounted in the Instron testing machine one at a time. 0.5 mm diameter round tip stainless-steel rod was fixed to the upper stage of the universal testing machine (Instron, Canton, MA, USA). The rod was centered over the canal orifice of each root. The universal testing machine (Instron) was adjusted and vertical compressive force was applied at a crosshead speed of 1mm/min. The Instron tester applied a slowly increasing force, at a rate of 1.0 mm per min, until the root fractured. This point was verified by the computer monitoring the Instron testing machine; at the same time the crack was heard, the monitor showed a sharp drop in force. The test was terminated at this point and the force applied was recorded. The maximum amount of force necessary to fracture every sample was recorded in Newton (N).

SECONDARY OUTCOMES:
Crack pattern | 2 minutes
  crack pattern is complete/incomplete

CONTACTS AND LOCATIONS:
Overall Officials: Farah Naz, BDS,FCPS, Study Director — Dow University of Health Sciences
Locations (1):
- Dow University of Health Sciences, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pawar AM, Pawar MG, Thakur B, Banga KS, Luke AM. Resistance to fracture of teeth instrumented using novel EndoStar E5 rotary versus ProTaper NEXT and WaveOne file systems. J Conserv Dent. 2018 Jan-Feb;21(1):52-56. doi: 10.4103/JCD.JCD_216_16. PMID 29628648
- [Background] Pawar AM, Barfiwala D, Pawar M, Metzger Z, Kfir A, Jain N. Assessment of the fracture resistance of teeth instrumented using 2 rotary and 2 reciprocating files versus the Self-Adjusting File (SAF): An ex vivo comparative study on mandibular premolars. J Conserv Dent. 2016 Mar-Apr;19(2):138-42. doi: 10.4103/0972-0707.178692. PMID 27099419
- [Background] Capar ID, Altunsoy M, Arslan H, Ertas H, Aydinbelge HA. Fracture strength of roots instrumented with self-adjusting file and the ProTaper rotary systems. J Endod. 2014 Apr;40(4):551-4. doi: 10.1016/j.joen.2013.08.030. Epub 2013 Oct 15. PMID 24666910
- [Background] Tavanafar S, Karimpour A, Karimpour H, Mohammed Saleh A, Hamed Saeed M. Effect of Different Instrumentation Techniques on Vertical Root Fracture Resistance of Endodontically Treated Teeth. J Dent (Shiraz). 2015 Mar;16(1 Suppl):50-5. PMID 26106635